CLINICAL TRIAL: NCT05677451
Title: A Double-blind, Randomized, Placebo-controlled Trial to Evaluate the Efficacy, Pharmacokinetics and Safety of Remibrutinib (LOU064) for 24 Weeks in Adolescents From 12 to Less Than 18 Years of Age With Chronic Spontaneous Urticaria Inadequately Controlled by H1-antihistamines Followed by an Optional Open-label Extension for up to Another 3 Years and an Optional Safety Long-term Treatment-free Follow-up Period for up to an Additional 3 Years
Brief Title: 24 Weeks Double-blind Randomized Placebo-controlled Trial to Evaluate Efficacy, PK, Safety of LOU064 in Adolescents (12 - <18) With CSU and Inadequate Response to H1-antihistamine Followed by Optional 3 Years Open-label Extension and an Optional 3 Years Safety Long-term Treatment-free Follow-up
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOU064F12301; 2022-502159-78-00 (Other: EU CT Number)
Record Dates: First submitted 2022-12-16; First posted 2023-01-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: BTK inhibitor; Chronic spontaneous urticaria; Urticaria activity score; Hives severity score; Itch severity score
MeSH Terms: conditions — Chronic Urticaria | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: LOU064 (blinded) (Experimental): LOU064 (blinded) taken orally b.i.d. for 24 weeks, followed by LOU064 (open-label) taken orally b.i.d. for up to 6 cycles of 24 weeks.
  Interventions: Drug: LOU064 (blinded)
- Arm 2: LOU064 placebo (blinded) (Placebo Comparator): LOU064 placebo (blinded) taken orally b.i.d. for 24 weeks (randomized in a 2:1 ratio arm 1: arm 2)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LOU064 (blinded) — LOU064 (blinded) active treatment
  Other Names: remibrutinib
  Arms: Arm 1: LOU064 (blinded)
Drug: placebo — matching active drug
  Arms: Arm 2: LOU064 placebo (blinded)

SUMMARY:
The purpose of this trial is:

1. to assess the efficacy, pharmacokinetics, and safety of remibrutinib vs. placebo in adolescents from 12 to < 18 years of age suffering from chronic spontaneous urticaria inadequately controlled by H1-antihistamines
2. to collect long-term efficacy, safety and tolerability data on remibrutinib in adolescents after having completed 24 weeks of treatment
3. to collect safety data in this population for up to three years after the last dose of study treatment

DETAILED DESCRIPTION:
This trial consists of 3 different periods:

1. the "core period", which is randomized and double-blind, during which 2/3 participants will receive remibrutinib and 1/3 will receive placebo for 24 weeks. Total duration: approximately 32 weeks (10 site visits).
2. an optional "open-label extension (OLE) period" proposed to all participants who completed 24 weeks of treatment of the "core period" and all scheduled assessments planned at week 24 visit . Depending on their CSU symptoms (as assessed by the doctor), participants will either receive remibrutinib for 24 weeks, or enter an observational treatment-free period for 1 year. If the CSU symptoms return during the observational period, the participants can switch to the treatment period at any time (decided by the doctor). At the end of the 24-week treatment period, if CSU is controlled, participants will enter the 1-year observational period, otherwise, they can continue with another cycle of 24-week remibrutinib treatment. The number of remibrutinib treatment or observational cycles will be limited to 6 times each. Total duration: from 1 year to approximately 3 years, and number of visits: from 3 to 15 (depending on the CSU symptoms).
3. an optional "long-term treatment-free follow-up period" proposed to all participants who completed at least 4 months treatment in the "OLE period". No treatment will be given. Duration: 3 years with 1 site visit and up to 4 phone call follow-up visits.

The primary clinical question of interest is what is the effect of remibrutinib treatment versus placebo on the change from baseline in UAS7, ISS7 and HSS7 scores after 12 weeks of treatment

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female adolescent participants aged >= 12 to < 18 years of age at the time of signing the informed consent
* CSU duration for >= 6 months prior to screening (defined as the onset of CSU determined by the investigator based on all available supporting documentation)
* Diagnosis of CSU inadequately controlled by second-generation H1-AH at the time of randomization defined as:
* The presence of itch and hives for ≥ 6 consecutive weeks prior to screening despite the use of second-generation H1-AH during this time period according to local treatment guidelines
* UAS7 score (range 0 - 42) >= 16, ISS7 score (range 0 - 21) >= 6 and HSS7 score (range 0 - 21) >= 6 during the 7 days prior to randomization (Day 1)
* Documentation of hives within three months before randomization (either at screening and/or at randomization; or documented in the participants' medical history)

Key Exclusion criteria:

* Previous use of remibrutinib or other BTK inhibitors
* Significant bleeding risk or coagulation disorders
* History of gastrointestinal bleeding
* Requirement for anti-platelet medication, except for acetylsalicylic acid up to 100 mg/d or clopidogrel up to 75 mg/d. The use of dual anti-platelet therapy (e.g., acetylsalicylic acid + clopidogrel) is prohibited
* History or current hepatic disease
* Evidence of clinically significant cardiovascular, neurological, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, hematological disorders, gastrointestinal disease or immunodeficiency that, in the investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant
* History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes
* Participants having a clearly defined predominant or sole trigger of their chronic urticaria (chronic inducible urticaria) including urticaria factitia (symptomatic dermographism), cold-, heat-, solar-, pressure-, delayed pressure-, aquagenic-, cholinergic-, or contact-urticaria
* Other diseases with symptoms of urticaria or angioedema, including but not limited to urticaria vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary angioedema, or drug-induced urticaria
* Any other skin disease associated with chronic itching that might influence in the investigator's opinion the study evaluations and results, e.g., atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus or psoriasis

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2032-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in UAS7 | Baseline, week 12
  The Urticaria Activity Score (UAS) is sum of the Hive Severity Score (HSS) and the Itch Severity Score (ISS). UAS7 is sum of the HSS7 and the ISS7 scores. Possible range of weekly UAS7 score is 0 to 42. Complete UAS7 response is UAS7 = 0.
  Negative change from baseline indicates improvement.
Change fron baseline in ISS7 | Baseline, Week 12
  Itch Severity Score (ISS) scale is 0 to 3. Score (ISS7) is derived by adding up average daily scores of 7 days preceding visit. Possible range of weekly score is therefore 0 to 21. Itch Severity Score scale: 0 - None 1 - Mild (minimal awareness, easily tolerated) 2 - Moderate (definite awareness, bothersome but tolerable) 3 - Severe (difficult to tolerate).
  Negative change from baseline indicates improvement.
Change from baseline in HSS7 | Baseline, Week 12
  Hives Severity Score (HSS) scale is 0 to 3. A weekly score (HSS7) is derived by adding up the average daily scores of the 7 days preceding the visit. Possible range of the weekly score is therefore 0 to 21. Hives Severity Score scale: 0 - None 1 - Mild (1-6 hives/12 hours) 2 - Moderate (7-12 hives/12 hours) 3 - Severe (>12 hives/12 hours).
  Negative change from baseline indicates improvement.

SECONDARY OUTCOMES:
Cmax of remibrutinib | At Week 12, before study drug intake, then after 30 min, 1 h, 2h, 3h and 4 h after study drug intake
  The maximum (peak) observed blood drug concentration after single dose administration
Tmax of remibrutinib | At Week 12, before study drug intake, then after 30 min, 1 h, 2h, 3h and 4 h after study drug intake
  The time to reach maximum (peak) blood drug concentration after single dose administration
AUClast of remibrutinib | At Week 12, before study drug intake, then after 30 min, 1 h, 2h, 3h and 4 h after study drug intake
  The Area Under the Curve (AUC) from pre-dose to the last measurable concentration sampling time
Absolute change from baseline in ISS7 | Baseline - Week 12
  Itch Severity Score (ISS) scale is 0 to 3. Score (ISS7) is derived by adding up average daily scores of 7 days preceding visit. Possible range of weekly score is therefore 0 to 21. Itch Severity Score scale: 0 - None 1 - Mild (minimal awareness, easily tolerated) 2 - Moderate (definite awareness, bothersome but tolerable) 3 - Severe (difficult to tolerate).
  Negative change from baseline indicates improvement.
Absolute change from baseline in HSS7 | Baseline - Week 12
  Hives Severity Score (HSS) scale is 0 to 3. A weekly score (HSS7) is derived by adding up the average daily scores of the 7 days preceding the visit. Possible range of the weekly score is therefore 0 to 21. Hives Severity Score scale: 0 - None 1 - Mild (1-6 hives/12 hours) 2 - Moderate (7-12 hives/12 hours) 3 - Severe (>12 hives/12 hours).
  Negative change from baseline indicates improvement.
Achievement of UAS7 ≤ 6 (yes/no) | Week 12 and over time
  Disease activity control is defined as UAS7 ≤ 6. The Urticaria Activity Score (UAS) is sum of the Hive Severity Score (HSS) and the Itch Severity Score (ISS). UAS7 is sum of the HSS7 and the ISS7 scores. Possible range of weekly UAS7 score is 0 to 42.
Achievement of UAS7 = 0 (yes/no) | Week 12 and over time
  Complete absence of hives and itch is defined as UAS7 = 0. The Urticaria Activity Score (UAS) is sum of the Hive Severity Score (HSS) and the Itch Severity Score (ISS). UAS7 is sum of the HSS7 and the ISS7 scores. Possible range of weekly UAS7 score is 0 to 42.
Absolute change from baseline in CDLQI score | Week 12
  The Children Dermatology life Quality Index (CDLQI) score range is 0 to 30, with 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Number of weeks without angioedema, assessed by the cumulative number of weeks with an AAS7 = 0 response | baseline - Week 12
  Angioedema Activity Score (AAS7) is a measure of the frequency and intensity of angioedema episodes. The total possible range of scores over 7 days is 0-105 where higher scores indicate increased angioedema activity.
Occurrence of treatment-emergent adverse events (AE) and serious adverse events (SAE) during the core period | 28 weeks
  To demonstrate the safety and tolerability of remibrutinib by assessing occurrence of treatment emergent adverse events and serious adverse events during the core period of the study.
Occurrence of treatment emergent AEs, and SAEs during the Open Label Extension (OLE) period | 3 years
  To demonstrate the safety and tolerability of remibrutinib by assessing occurrence of treatment emergent adverse events and serious adverse events during the OLE period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- United States (12):
  - Kern Research, Bakersfield, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Pediatric Dermatology of Miami at the Pediatric CoE, Coral Gables, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Endeavor Health, Glenview, Illinois
  - Allergy and Asthma Specialist P S C, Owensboro, Kentucky
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Allergy Asthma and Clinical Research, Oklahoma City, Oklahoma
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - RFSA Dermatology, San Antonio, Texas
  - Allergy Associates of Utah, Sandy City, Utah
  - Seattle Allergy and Asthma Rsch, Seattle, Washington
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Santiago, Chile
- China (3):
  - Novartis Investigative Site, Guangdong, Guangzhou
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
- Germany (5):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Pokfulam
- Italy (7):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Bari
  - Novartis Investigative Site, Napoli
- Japan (5):
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kamimashi-gun, Kumamoto
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Itabashi-ku, Tokyo
- Novartis Investigative Site, Kuching, Sarawak, Malaysia
- Netherlands (2):
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Utrecht
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Singapore, Singapore
- South Africa (2):
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, Cape Town, Western Cape
- Spain (3):
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
- Thailand (2):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
- United Kingdom (3):
  - Novartis Investigative Site, Peterborough, Cambridgeshire
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com